CLINICAL TRIAL: NCT06291012
Title: Evaluation of a Therapeutic Strategy to Reduce the Duration of Antibiotic Therapy for Community-acquired Alveolar Pneumonia in Children: a Randomized Controlled Non-inferiority Trial
Brief Title: Stopping Pneumonia Antibiotherapy Regimen Early
Acronym: SPARE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL22_0399; 2024-512236-30-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Community-acquired Pneumonia; Child, Only
Keywords: Antibiotics management; Amoxicillin
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: The randomization will be carried out by minimization with stratification on the investigating center and age (< 1 year and ≥ 1 year)
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short arm (Experimental): Antibiotic therapy for 3 to 5 days depending on response
  Interventions: Drug: Quick response: Amoxicillin for 3 days; Drug: Delayed response: Amoxicillin for 5 days
- Long arm (Active Comparator): Antibiotic therapy for 5 to 7 days depending on response
  Interventions: Drug: Quick response: Amoxicillin for 5 days; Drug: Delayed response: Amoxicillin for 7 days

INTERVENTIONS:
Drug: Quick response: Amoxicillin for 3 days — Once the diagnosis of community-acquired alveolar pneumonia has been made, the investigator taking charge of the child writes a prescription for amoxicillin at a dosage of 80-100 mg/kg/day in 3 oral doses (morning, noon and evening), for a period of 4 days, before delivery of treatment to the family. The investigator will carry out a clinical re-evaluation on day 3 (D3), during which he will decide on the final duration of treatment.
  In case of rapid response*: Immediate stop of antibiotherapy (after 9 complete doses)
  *A rapid response is determined by a favorable clinical evolution (MASCOT 2002 study)
  Other Names: Quick response (3 days)
  Arms: Short arm
Drug: Delayed response: Amoxicillin for 5 days — Once the diagnosis of community-acquired alveolar pneumonia has been made, the investigator taking charge of the child writes a prescription for amoxicillin at a dosage of 80-100 mg/kg/day in 3 oral doses (morning, noon and evening), for a period of 4 days, before delivery of treatment to the family. The investigator will carry out a clinical re-evaluation on day 3 (D3), during which he will decide on the final duration of treatment.
  In case of delayed response: Continuation of antibiotic therapy for up to 5 days
  Other Names: Delayed response (5 days)
  Arms: Short arm
Drug: Quick response: Amoxicillin for 5 days — Once the diagnosis of community-acquired alveolar pneumonia has been made, the investigator taking charge of the child writes a prescription for amoxicillin at a dosage of 80-100 mg/kg/day in 3 oral doses (morning, noon and evening), for a period of 4 days, before delivery of treatment to the family. The investigator will carry out a clinical re-evaluation on day 3 (D3), during which he will decide on the final duration of treatment.
  In case of rapid response*: Continuation of antibiotherapy for up to 5 days
  *A rapid response is determined by a favorable clinical evolution (MASCOT 2002 study)
  Other Names: Quick response (5 days)
  Arms: Long arm
Drug: Delayed response: Amoxicillin for 7 days — Once the diagnosis of community-acquired alveolar pneumonia has been made, the investigator taking charge of the child writes a prescription for amoxicillin at a dosage of 80-100 mg/kg/day in 3 oral doses (morning, noon and evening), for a period of 4 days, before delivery of treatment to the family. The investigator will carry out a clinical re-evaluation on day 3 (D3), during which he will decide on the final duration of treatment.
  In case of delayed response: Continuation of antibiotic therapy for up to 7 days
  Other Names: Delayed response (7 days)
  Arms: Long arm

SUMMARY:
The hypothesis for this trial is that an antibiotic strategy for the management of non-severe community-acquired alveolar pneumonia in children aged 3 to 59 months, including amoxicillin 80-100 mg/kg/day for at least 3 days in case of rapid response and 5 days in case of delayed response, would not be inferior to current French recommendations (antibiotic therapy for 5 days in case of rapid response and 7 days in case of delayed response) in terms of treatment of failure rate at 7 days.

DETAILED DESCRIPTION:
Introduction:

The World Health Organization (WHO) has declared antimicrobial resistance to be one of the 10 greatest threats to public health. As such, it has issued recommendations for children for the diagnosis and treatment of pneumonia with amoxicillin for 3 days. However, this strategy includes viral infections and therefore cannot be extrapolated directly to countries with a high level of access to healthcare, where the aim is to treat only bacterial pneumonia and for the shortest possible time to limit the emergence of resistant bacteria. Thus, our study proposes to use a definition of pneumonia adapted to countries with a high level of access to healthcare and to test an adaptive treatment regimen including a clinical reassessment at D3, which will propose a treatment limited to 3 days in case of rapid response and 5 days in case of delayed response.

Aim:

The aim of this trial is to demonstrate the non-inferiority of a strategy of antibiotic treatment with amoxicillin 80-100 mg/kg/day for 3 days in the case of a rapid response or 5 days in the case of a delayed response, versus antibiotic treatment for 5 days in the case of a rapid response or 7 days in the case of a delayed response for the management of non-severe community-acquired alveolar pneumonia in children between 3 and 59 months, in terms of the rate of treatment failure at 7 days.

Methods:

As the hypothesis is not that a shorter antibiotic regimen is more effective in this indication, a non-inferiority trial is the most appropriate design to assess whether this efficacy is broadly comparable with the reference regimen. The primary endpoint chosen is the one already used in an international clinical trial on this disease in children, which has been agreed upon.

In order to meet the objective of the study, 1100 patients will be included.

* At D0, patients will be included and randomized by the investigator, and will begin their treatment: Short arm: treatment by amoxicillin 80-100 mg/kg/d for 3 days if rapid response or 5 days if delayed response; or Long arm: treatment by amoxicillin 80-100 mg/kg/d for 5 days if rapid response or 7 days if delayed response. A prescription and follow-up diary will be given to the family.
* At D3, the doctor will assess the response to the treatment. If the response is assessed as rapid, then the investigator will reduce the duration of antibiotic treatment depending on the arm to which the child has been randomized. Parents will continue to complete the follow-up diary until D7.
* At the D7 visit, the investigator evaluates the primary endpoint and some of the secondary endpoints.
* At the D30 visit, the investigator assesses of last secondary endpoints.

Given the non-inferiority design, data will be analyzed on a per protocol basis for the primary analysis. The per-protocol population will be defined by radiologist of pneumonia diagnosis, at least one dose of amoxicillin, and having primary endpoint assessment data at 7 days. Non-inferiority will be declared if the lower bound of the confidence interval of the difference in failure rate between the 3-day and 5-day arms is less than 3.5%.

ELIGIBILITY:
Inclusion Criteria:

* Child with a diagnosis of community-acquired alveolar pneumonia defined as an association of 3 major criteria + at least 3/5 minor criteria:

  * Major criteria: Fever (> 38°C), Polypnea and Chest x-ray
  * Minor criteria: Localized crackles, C-Reactive Protein (CRP) > 80mg/L, Alteration of general condition, Cough and Pulmonary condensation syndrome.
* Child with an episode that began less than 7 days before inclusion, in the community.
* Absence of hospitalization criteria

Exclusion Criteria:

* Pre-existing underlying pathology: acquired or hereditary immune deficiencies, cardiac pathologies, chronic respiratory failure or pulmonary malformations, neurological or muscular diseases at risk of respiratory decompensation, serious chronic kidney diseases and nephrotic syndromes, sickle cell anemia, diabetes, chronic liver diseases, oncological pathologies and hematological, organ and hematopoietic stem cell transplants, inflammatory and/or autoimmune diseases receiving immunosuppressive treatment, people infected with HIV, obese people with a body mass index (BMI) ≥ the 97th percentile
* Asthma with basic treatment
* Wheezing during the episode
* Presence of pleural effusion on radiography
* Presence of toxin signs
* Antibiotic therapy within 48 hours before inclusion
* Anti-inflammatory therapy within 48 hours before inclusion
* Allergy or contraindication to penicillin
* History of more than 2 bacterial pneumonias per year
* Associated infection requiring more than 3 days of antibiotics
* Patient hospitalized within 15 days before inclusion
* Failure to obtain informed consent by the legal representative(s)
* Patient whose legal representatives are unable to read/write french language
* Patient not affiliated with or not benefiting from a national health insurance scheme
* Patient participating in another interventional research involving human person

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic failure rate D7 | Day 7
  Day 0 (D0) is defined as the 1st day of taking amoxicillin.
  The rate of therapeutic failure on day 7 (D7) defined by:
  * A change in antibiotherapy necessary before D7 due to a lack of satisfactory clinical response or clinical deterioration of the pneumonia.
  * A decision to resume or continue antibiotic therapy after D7 in connection with the pneumonia.
  * Hospitalization or death due to clinical deterioration related to community-acquired pneumonia.
  This definition is based on that already used in a clinical trial carried out in Israel (6. Greenberg D, Givon-Lavi N, Sadaka Y, Ben-Shimol S, Bar-Ziv J, Dagan R. Short-course Antibiotic Treatment for Community-acquired Alveolar Pneumonia in Ambulatory Children. Pediatr Infect Dis J. 2014 Feb;33(2):136-42).

SECONDARY OUTCOMES:
Therapeutic failure rate on D30 | Day 30
  Day 0 (D0) is defined as the 1st day of taking amoxicillin.
  Therapeutic failure 30 days after , defined by:
  * The occurrence of hospitalization linked to the initial episode.
  * An abnormal check-up chest x-ray at 1 month with persistent pneumonia.
  * The occurrence of complications of pneumonia (severe sepsis, pleurisy, pulmonary sequelae).
  * Relapse, defined by the development of signs of pneumonia 6 to 14 days after the respiratory rate returns to normal.
Adverse effects | Day 0, Day 3, Day 7 and Day 30
  Occurrence of adverse effects attributable to antibiotics during and after taking amoxicillin.
  Day 0 (D0) is defined as the 1st day of taking amoxicillin.
Compliance | Day 7, or Day 30 in case of therapeutic failure
  Compliance is recorded in a monitoring log, completed by the child's family, throughout the duration of antibiotic therapy.
  Day 0 (D0) is defined as the 1st day of taking amoxicillin.
Duration of antibiotic therapy | Day 7 and Day 30
  The duration of antibiotic therapy is collected in a monitoring log completed by the patients' families, and during the interview at visits on D7 and D30.
  Day 0 (D0) is defined as the 1st day of taking amoxicillin.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah DUTRON, MD, Study Director — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haider BA, Saeed MA, Bhutta ZA. Short-course versus long-course antibiotic therapy for non-severe community-acquired pneumonia in children aged 2 months to 59 months. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD005976. doi: 10.1002/14651858.CD005976.pub2. PMID 18425930
- [Background] Pakistan Multicentre Amoxycillin Short Course Therapy (MASCOT) pneumonia study group. Clinical efficacy of 3 days versus 5 days of oral amoxicillin for treatment of childhood pneumonia: a multicentre double-blind trial. Lancet. 2002 Sep 14;360(9336):835-41. doi: 10.1016/S0140-6736(02)09994-4. PMID 12243918
- [Background] Ginsburg AS, Mvalo T, Nkwopara E, McCollum ED, Phiri M, Schmicker R, Hwang J, Ndamala CB, Phiri A, Lufesi N, May S. Amoxicillin for 3 or 5 Days for Chest-Indrawing Pneumonia in Malawian Children. N Engl J Med. 2020 Jul 2;383(1):13-23. doi: 10.1056/NEJMoa1912400. PMID 32609979
- [Background] Chang AB, Grimwood K. Antibiotics for Childhood Pneumonia - Do We Really Know How Long to Treat? N Engl J Med. 2020 Jul 2;383(1):77-79. doi: 10.1056/NEJMe2016328. No abstract available. PMID 32609987
- [Background] Greenberg D, Givon-Lavi N, Sadaka Y, Ben-Shimol S, Bar-Ziv J, Dagan R. Short-course antibiotic treatment for community-acquired alveolar pneumonia in ambulatory children: a double-blind, randomized, placebo-controlled trial. Pediatr Infect Dis J. 2014 Feb;33(2):136-42. doi: 10.1097/INF.0000000000000023. PMID 23989106
- [Background] Cohen R, Angoulvant F, Biscardi S, Madhi F, Dubos F, Gillet Y. Antibiotic treatment of lower respiratory tract infections. Arch Pediatr. 2017 Dec;24(12S):S17-S21. doi: 10.1016/S0929-693X(17)30513-4. PMID 29290229
- [Background] Gauzit R, Castan B, Bonnet E, Bru JP, Cohen R, Diamantis S, Faye A, Hitoto H, Issa N, Lebeaux D, Lesprit P, Maulin L, Poitrenaud D, Raymond J, Strady C, Varon E, Verdon R, Vuotto F, Welker Y, Stahl JP. Anti-infectious treatment duration: The SPILF and GPIP French guidelines and recommendations. Infect Dis Now. 2021 Mar;51(2):114-139. doi: 10.1016/j.idnow.2020.12.001. Epub 2020 Dec 31. No abstract available. PMID 34158156
- [Background] Same RG, Amoah J, Hsu AJ, Hersh AL, Sklansky DJ, Cosgrove SE, Tamma PD. The Association of Antibiotic Duration With Successful Treatment of Community-Acquired Pneumonia in Children. J Pediatric Infect Dis Soc. 2021 Apr 3;10(3):267-273. doi: 10.1093/jpids/piaa055. PMID 32525203
- [Background] Leekha S, Terrell CL, Edson RS. General principles of antimicrobial therapy. Mayo Clin Proc. 2011 Feb;86(2):156-67. doi: 10.4065/mcp.2010.0639. PMID 21282489
- [Background] Angoulvant F, Cohen R, Doit C, Elbez A, Werner A, Bechet S, Bonacorsi S, Varon E, Levy C. Trends in antibiotic resistance of Streptococcus pneumoniae and Haemophilus influenzae isolated from nasopharyngeal flora in children with acute otitis media in France before and after 13 valent pneumococcal conjugate vaccine introduction. BMC Infect Dis. 2015 Jun 21;15:236. doi: 10.1186/s12879-015-0978-9. PMID 26093673
- [Background] Angoulvant F, Levy C, Grimprel E, Varon E, Lorrot M, Biscardi S, Minodier P, Dommergues MA, Hees L, Gillet Y, Craiu I, Zenkhri F, Dubos F, Guen CG, Launay E, Martinot A, Cohen R. Early impact of 13-valent pneumococcal conjugate vaccine on community-acquired pneumonia in children. Clin Infect Dis. 2014 Apr;58(7):918-24. doi: 10.1093/cid/ciu006. Epub 2014 Feb 13. PMID 24532543
- See also: WHO declared antimicrobial resistance one of the 10 biggest public health threats facing humanity — https://www.who.int/fr/news-room/fact-sheets/detail/pneumonia
- See also: ANSM: All committed to better use of antibiotics (2021, November) — https://ansm.sante.fr/actualites/tous-engages-pour-un-meilleur-usage-des-antibiotiques
- See also: Review on antimicrobial resistance. Tackling drug-resistant infections globally: Final report and recommendations. (2016 May) — https://amr-review.org/sites/default/files/160518_Final%20paper_with%20cover.pdf
- See also: General principles and advice for prescribing antibiotics as a first resort (2014, February) — https://www.has-sante.fr/upload/docs/application/pdf/2014-02/conseils_prescription_antibiotiques_rapport_d_elaboration.pdf